CLINICAL TRIAL: NCT06927947
Title: Testing Effectiveness of Navigation Interventions to Increase Uptake of Cascade Genetic Testing Among Relatives of Individuals Diagnosed With Hereditary Cancer Syndromes
Brief Title: Navigation Interventions to Improve Cascade Genetic Testing Among Relatives of Patients With Hereditary Cancer Syndromes
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: UMCC 2024.087; NCI-2025-02246 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); HUM00257832 (Other: University of Michigan)
Record Dates: First submitted 2025-04-04; First posted 2025-04-15 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-10

CONDITIONS: Hereditary Malignant Neoplasm; Hereditary Neoplastic Syndrome
MeSH Terms: conditions — Neoplastic Syndromes, Hereditary | interventions — Health Promotion; Educational Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prevention (Cascade Genetic Testing Platform) (Experimental): PROBANDS: Probands use the relative invitation tool to invite at-risk relatives to participate.
  RELATIVES: Participants receive access to the virtual Cascade Genetic Testing Platform, which includes a Genetic Testing Family Letter and access to the VGN. The Genetic Testing Family Letter provides information about the genetic diagnosis in the family, instructions for the relatives on how to schedule a genetic evaluation, and contact information for the U-M Cancer Genetics Clinic. The VGN is an interactive web-based tool that provides personalized information addressing readiness, barriers and motivators to testing, and knowledge, and presents educational content about genetic testing and information about testing options, including how to access them on study.
  Interventions: Other: Communication Intervention; Other: Health Promotion and Education; Other: Informational Intervention; Other: Survey Administration

INTERVENTIONS:
Other: Communication Intervention — Use relative invitation tool
Other: Health Promotion and Education — Receive access to the VGN
Other: Informational Intervention — Receive access to a Genetic Testing Family Letter
Other: Survey Administration — Ancillary studies

SUMMARY:
This clinical trial tests whether various web-based tools can help improve communication about hereditary cancer risk in families and decrease barriers to genetic testing for relatives of patients with hereditary cancer syndromes. Between 5% and 10% of all cancers are caused by genetic changes that are hereditary, which means that they run in families. Some kinds of cancer or certain cancers diagnosed in biological relatives may mean patients are more likely to have a genetic change. Once a genetic change is identified in a family, other biological relatives can choose to undergo testing themselves to better understand their cancer risk. The uptake of genetic testing in other biological relatives once a genetic condition is identified is about 20% to 30%. The Cascade Genetic Testing Platform is a virtual tool that seeks to overcome barriers related to logistics of family communication and improve dissemination of genetic testing information which is clinically actionable for individuals at highest risk for cancer. Using the Cascade Genetic Testing Platform may improve ways to share information about hereditary risk with biological relatives.

DETAILED DESCRIPTION:
03JUN2025- Amendment was approved that shorten the study timeline from 12 to 6 months. We believe this is sufficient to capture our primary outcome (participation) and a shorter timeline may keep participants more engaged.

ELIGIBILITY:
Inclusion Criteria:

* PROBANDS: Clinically confirmed autosomal dominant pathogenic germline variant (PGV) associated with a hereditary cancer syndrome
* PROBANDS: Previous evaluation by the University of Michigan (U-M) Cancer Genetics Clinic
* PROBANDS: ≥ 18 years old
* PROBANDS: Able to speak and read English
* PROBANDS: Access to the internet
* RELATIVES: Biological relative of proband
* RELATIVES: ≥ 18 years old
* RELATIVES: Able to speak and read English
* RELATIVES: Access to the internet
* RELATIVES: Have not completed germline genetic testing, per self-report at baseline

Exclusion Criteria:

* RELATIVES: Prior clinical germline genetic testing for cancer or already have an upcoming appointment scheduled with a genetics provider, per self-report at baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2025-09-23 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of probands that utilize the invitation tool | Up to 6 Months
  Will be defined as inviting at least 1 eligible at-risk relative. Will be assessed using descriptive statistics. Will be tabulated and summarized. Continuous variables will be summarized by mean, median, and standard deviation; histograms and boxplots will be used to further assess distributional characteristics of these variables. Categorical variables will be tabulated with frequencies and percentages. Will be estimated and presented along with a 95% confidence interval.
Percentage of invited relatives that engage | Up to 6 Months
  Will be defined as enrolling in the study and accessing the informational content (letter and/or virtual genetics navigator) at least 1 time. Will be assessed using descriptive statistics. Will be tabulated and summarized. Continuous variables will be summarized by mean, median, and standard deviation; histograms and boxplots will be used to further assess distributional characteristics of these variables. Categorical variables will be tabulated with frequencies and percentages. Will be estimated and presented along with a 95% confidence interval.

SECONDARY OUTCOMES:
Extent of utilization of the invitation portal by probands | Up to 6 Months
  Will be measured by the number of relatives invited out of the estimated number of eligible at-risk relatives (e.g. blood-related, have not completed genetic testing, living, 18 years or older). Will be calculated based on previously collected family records as reviewed by a genetic counselor, in conjunction with any updated information received from participants. Will be assessed using descriptive statistics. Will be tabulated and summarized. Continuous variables will be summarized by mean, median, and standard deviation; histograms and boxplots will be used to further assess distributional characteristics of these variables. Categorical variables will be tabulated with frequencies and percentages. Will be estimated and presented along with a 95% confidence interval.
Percentage of relatives invited who subsequently enroll in the study | Up to 6 Months
  Will be assessed using descriptive statistics. Will be tabulated and summarized. Continuous variables will be summarized by mean, median, and standard deviation; histograms and boxplots will be used to further assess distributional characteristics of these variables. Categorical variables will be tabulated with frequencies and percentages. Will be estimated and presented along with a 95% confidence interval.
Percentage of relative participants who have either scheduled or completed genetic testing | Up to 3 months
  Will be assessed using descriptive statistics. Will be tabulated and summarized. Continuous variables will be summarized by mean, median, and standard deviation; histograms and boxplots will be used to further assess distributional characteristics of these variables. Categorical variables will be tabulated with frequencies and percentages. Will be estimated and presented along with a 95% confidence interval.

CONTACTS AND LOCATIONS:
Overall Officials: Elena M Stoffel, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No